CLINICAL TRIAL: NCT01344603
Title: Epidural Analgesia in Cardiac Surgery
Brief Title: Epidural and Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Landoni Giovanni, Vita-Salute University of Milano, Italy
Other Study IDs: HSR epi CCH 38
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Cardiac Disease
Keywords: cardiac surgery; cardiac anesthesia; epidural
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- epidural
- standard

SUMMARY:
In the present study the investigators test the hypothesis that the epidural anesthesia added on the general anesthesia is able to improve patient's outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery
* adult (>18y)
* sternotomy

Exclusion Criteria:

* abnormal coagulation profile
* antiplatelet medications (other than aspirin)
* ongoing anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing cardiac surgery
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Università Vita-Salute San Raffaele, Milan, MI, Italy